CLINICAL TRIAL: NCT04030091
Title: Pilot Study for Evaluation of the Impact of Pulsatile Insulin Infusion Therapy on Vascular Function in Patients With Type 1 and Type 2 Diabetes Mellitus
Brief Title: Pulsatile Insulin Infusion Therapy in Patients With Type 1 and Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sciema UG (Other)
Collaborators: Innovative Diabetes Treatment Studies LLC. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DCTI-PIT-001
Record Dates: First submitted 2019-07-15; First posted 2019-07-23 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1 | interventions — Insulin

STUDY DESIGN:
Intervention Model Description: 1 arm of 2 hours pulsatile insulin infusion treatment vs. a second arm of 3 hours pulsatile insulin infusion treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3 hour pulsatile normal insulin infusion treatment (Experimental): the pulsatile insulin infusion treatment will be applied for 3 hours once a week with 10 pulses of 3 U of humulin R 100 IU/mL insulin per hour
  Interventions: Drug: 3 hours humulin R 100 IU/mL PIT
- 2 hour pulsatile normal insulin infusion treatment (Experimental): the pulsatile insulin infusion treatment will be applied for 2 hours once a week with 10 pulses of 3 U of humulin R 100 IU/mL insulin per hour
  Interventions: Drug: 2 hours humulin R 100 IU/mL PIT

INTERVENTIONS:
Drug: 3 hours humulin R 100 IU/mL PIT — PIT procedure: a venous catheter will be placed into one superficial vein at one arm, which will be connected to the insulin infusion pump and a glucose infusion pump via a three-way connector. Endothelial function will be measured by means of the Vendys 2 device. The blood glucose will be tested by means of a POCT meter and the CGM, and the PIT procedure will be started (10 pulses of 3 U of regular human insulin per hour). Blood glucose will be tested every 5 to 10 min and glucose infusion will be started once a drop in blood glucose is detected. Adjustment of glucose administration will be performed until a stable glucose value between 80 mg/dL to 160 mg/dL is reached. In parallel, endothelial function will be measured every 30 min. At the end of the PIT procedure, the venous catheter will be removed and the patient will be discharged until the next visit.
  Arms: 3 hour pulsatile normal insulin infusion treatment
Drug: 2 hours humulin R 100 IU/mL PIT — As described for the Intervention "3 hours of pulsatile insulin infusion (PIT) with humulin R 100 IU/mL", the treatment duration is just one hour less.
  Arms: 2 hour pulsatile normal insulin infusion treatment

SUMMARY:
This study is an open label, prospective, randomised comparative, single center study. In the present study, the impact of a 12-week pulsatile insulin infusion therapy (PIT) with Humulin R 100 from

DETAILED DESCRIPTION:
During the screening visit the patient will arrive at the study site and written informed consent will be obtained. Inclusion and exclusion criteria will be controlled and blood will be drawn for HbA1c and safety parameters. A point of care treatment (POCT) pregnancy test will be conducted in women of childbearing age. Patient demographics and history will be collected and a physical examination will be performed. The patient will complete a QoL, the continous glucose monitoring (CGM) sensor will be placed and trained, and the schedules for the subsequent treatment visits will be made. Also, the randomization (2 h vs 3 h) will be performed.

During the initiation visit , a series of clinical assessments will be made to document the patient status with respect to secondary complications: sensory nerve perception thresholds (tuning fork and path tester), retinopathy (RetinaVue camera). An ECG will be conducted, and blood will be drawn for assessment of the efficacy parameters. Thereafter the pulsatile insulin infusion therapy (PIT) procedure will be initiated.

For each PIT procedure: a venous catheter will be placed into one superficial vein at one arm, which will be connected to the insulin infusion pump and a glucose infusion pump via a three-way connector. Endothelial function will be measured by means of the Vendys 2 device (manufacturer: endothelix). The blood glucose will be tested by means of a POCT meter and the CGM, and the PIT procedure will be started (10 pulses of 3 U of regular human insulin per hour). Blood glucose will be tested every 5 to 10 min and glucose infusion will be started once a drop in blood glucose is detected. Adjustment of glucose administration will be performed until a stable glucose value between 80 mg/dL to 160 mg/dL is reached. In parallel, endothelial function will be measured every 30 min. At the end of the PIT procedure, the venous catheter will be removed and the patient will be discharged until the next visit.

During all consecutive treatment visits the patient will arrive at the investigational site at the agreed time-point and information regarding potential adverse events will be collected. Vital signs will be measured and the PIT procedure will be performed as described. At visits V6 and V10 additional examinations (assessments of neuropathy and retinopathy, blood draws for efficacy parameters, diabetes treatment satifaction questionnaire (DTSQ) questionnaire) will be performed.

During the final Visit the assessments from baseline (ECG, physical examination, neuropathy assessments, retinopathy assessment, blood draws for all safety and efficacy parameters incl. messenger ribonucleic acid (mRNA) analysis) will be repeated. The patient will complete a final DTSQ questionnaire, which concludes the participation in the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained prior to any trial-related activities
2. Male or female > 18 years
3. Diagnosed with Type 1 or 2 Diabetes ≥ 2 years
4. HbA1c <10%
5. Nephropathy with GFR between 30 and 60 mL/min/1,73m2 or < 75 GFR together with proteinuria and/or elevated creatinine levels
6. Patient is naïve to pulsatile insulin treatment

Exclusion Criteria:

1. Patients participating in another investigational drug study
2. Current or history of dialysis therapy
3. Anemia with hemoglobin < 10 g/dL
4. Unstable significant cardiovascular disease with admission to emergency room or hospital in last 45 days
5. Patients with diagnosed renal failure from non-diabetic etiology
6. Pregnancy or breast feeding
7. Patient unwillingness to use a CGM device, or inability (with or without family assistance) to replace the sensor every two weeks on the study CGM device
8. Drug or alcohol abuse
9. Sexually active woman of childbearing age not practicing birth control by accepted methods
10. Lack of compliance or other reason that in the discretion of the investigator precludes satisfactory participation in the study
11. Any severe illness preventing participation in the study per protocol (in the discretion of the investigator)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-09-06 (Actual); Primary Completion 2020-10-19 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Endothelial function | 1 hour
  Impact of PIT on endothelial function before and one hour after the PIT initiation measured with the Vendys2 device

SECONDARY OUTCOMES:
Renal function | 13 weeks
  It will be assessed whether insulin resistance has improved or worsened over the course of the study.
  Measured laboratory parameters for renal function (GFR, creatinine, proteinurea)
nerve function | 13 weeks
  Sensory nerve function (pathtester, tuning fork). It will be assessed whether insulin resistance has improved or worsened over the course of the study.
Retinopathy | 13 weeks
  Retinopathy will be measured with the RetinaVue device. It will be assessed whether Retinopathy has improved or worsened over the course of the study.
HbA1c | 13 weeks
  metabolic control
Insulin resistance | 13 weeks
  For assessment of insulin resistance glucose, retinol-binding protein 4 (RBP4), angiopoetin2, adiponectin, interleukin 6 (IL-6), hsCRP, glucagon, insulin, c-peptide, and intact Proinsulin will be measured. Finally, it is assessed whether insulin resistance has improved or worsened over the course of the study.
Diabetes treatment satisfaction questionnaire | 13 weeks
  Eight questions about the patient´s satisfaction with the diabetes treatment. Answer possibilities range form 1 (very good) to 10 (very bad)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Pfuetzner, Prof. Dr. Dr., Principal Investigator — Pfützner Science & Health Institute GmbH
Locations (2):
- NYC Research, Inc., New York, New York, United States
- Pfützner Science & Health Institute GmbH, Mainz, Rhineland-Palatinate, Germany